CLINICAL TRIAL: NCT06845449
Title: Tenting Screws Combined With Particulate Autogenous and Xenogenic Bone Versus Autogenous Ring Block Grafts Combined With Xenogenic Bone During Horizontal Ridge Augmentation
Brief Title: Tenting Screws Versus Autogenous Ring Block Grafts During Horizontal Ridge Augmentation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 333
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Horizontal Ridge Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tenting screw group (Experimental)
  Interventions: Procedure: tenting screw combined with particulate autogenous
- non screw group (Active Comparator)
  Interventions: Procedure: autogenous ring block grafts combined with xenogenic bone

INTERVENTIONS:
Procedure: tenting screw combined with particulate autogenous — In Tenting screw cases, the screws will be placed in suitable positions and depths, blocks will be crushed into particulates which will then be mixed with equal amount of bovine particles. the mixture will be applied to the recipient site all around the tenting screws a resorbable collagen membrane (CM) will be shaped and placed over the graft and fixed using subperiosteal sutures.
  Arms: tenting screw group
Procedure: autogenous ring block grafts combined with xenogenic bone — In the non screw group, the blocks will be adapted to fit the recipient sites and secured to the alveolar bone using titanium bone fixation screws. Following the placement of the blocks, bovine particles will be applied over the graft and into any remaining gaps between the block and the recipient site, a resorbable collagen membrane (CM) will be shaped and placed over the graft and fixed using subperiosteal sutures
  Arms: non screw group

SUMMARY:
After administering local anesthesia,. A full-thickness mucoperiosteal flap will be incised and be reflected to expose the alveolar bone. The dimensions of the defect will be measured using a periodontal probe to determine the appropriate size of the block graft or the quantity of particle bone graft required.

In the non screw group, the blocks will be adapted to fit the recipient sites and secured to the alveolar bone using titanium bone fixation screws. Following the placement of the blocks, bovine particles will be applied over the graft and into any remaining gaps between the block and the recipient site, a resorbable collagen membrane (CM) will be shaped and placed over the graft and fixed using subperiosteal sutures.

In Tenting screw cases, the screws will be placed in suitable positions and depths, blocks will be crushed into particulates which will then be mixed with equal amount of bovine particles. the mixture will be applied to the recipient site all around the tenting screws a resorbable collagen membrane (CM) will be shaped and placed over the graft and fixed using subperiosteal sutures.

The flaps will then be sutured

ELIGIBILITY:
Inclusion Criteria:

* Patient has anterior maxillary horizontal defect less than 4mm in the alveolar ridge and (classified as class III or IV atrophy according to Cawood and Howell classification). (Cawood & Howell, 1988require horizontal bone augmentation in anterior maxilla before dental implant placement and in need of an implant-supported restoration in at least one site,
* Adult individuals aged 18 years or older
* Satisfactory oral hygiene,
* No previous history of bone augmentation procedures at the site to be treated in the study,
* The ability to comprehend and provide informed consent.

Exclusion Criteria:

* Uncontrolled systemic disorders,
* Prior irradiation in the head and neck region,
* Immunosuppression or compromised immune system,
* Oral disorders such as lichen planus, ongoing or recent treatment with intravenous amino- bisphosphonates, untreated periodontitis,
* Poor oral hygiene and motivation,
* Parafunctional habits, pregnancy or lactation,
* Substance abuse involving drugs or alcohol, psychiatric disorders, a history (within the last 3 months) of regular use of smokeless chewing tobacco, smoking a pipe, cigar, or more than 10 cigarettes per day, acute or chronic infection or inflammation in the area, or
* Extraction with less than 3 months of healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone width gain | 6months

CONTACTS AND LOCATIONS:
Locations (1):
- Nahda University, Beni-seuf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided